CLINICAL TRIAL: NCT06129318
Title: Investigation of the Effects of Pharmaceutical Care Provided by a Clinical Pharmacist on Stroke Patients
Brief Title: :Effects of Pharmaceutical Care in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Mesut Sancar, Prof. Dr., Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MUHSI-2020/08-34
Record Dates: First submitted 2023-10-19; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pharmacist Led Pharmaceutical Care (Experimental): In addition to usual care services, the intervention group was provided with pharmaceutical care by a clinical pharmacist.
  Interventions: Behavioral: Clinical Pharmacist Led Pharmaceutical Care
- Control Group (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Clinical Pharmacist Led Pharmaceutical Care — Within the scope of pharmaceutical care, medication review services for past and current medication use were provided by the clinical pharmacist. The patients in the intervention group were given verbal information about the definition of stroke, symptoms, how to manage risk factors, and their medications by the clinical pharmacist on the day of discharge, in addition to the neurologist. Each patient in the intervention group had a scheduled meeting with the clinical pharmacist. During the 1-year follow-up the patient education given by the clinical pharmacist was repeated every 3 months.
  Arms: Clinical Pharmacist Led Pharmaceutical Care

SUMMARY:
To evaluate the effects of the 1-year pharmaceutical care program offered by the clinical pharmacist to the patients admitted to the neurology service with the diagnosis of stroke, on medication adherence, quality of life, and clinical outcomes of the patients.

DETAILED DESCRIPTION:
The study was conducted as a parallel randomized controlled study in the Neurology Clinic of a University Hospital in Turkey. Patients were randomly assigned to intervention and usual care groups. While the patients in the usual care group are given routine health services by the neurologist during their hospitalization and for 1 year after discharge; In addition to these routine services, the intervention group was provided with pharmaceutical care by a clinical pharmacist during the same period. The study was always conducted by the same neurologist and clinical pharmacist. Patient medication adherence, quality of life, and clinical parameters were evaluated at the beginning of the study and at the 12th month.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with stroke,
* being 18 years old or older,
* being in the cognition to receive the training to be given

Exclusion Criteria:

* Not having adequate cognitive function such as dementia,
* being pregnant, lactating,
* having cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 1, 3, 6, 9 and 12 months
  Blood pressure was checked and recorded by a qualified nurse during the hospital stay and at control visits. Measurements were recorded as mmHg.
Medication Adherence | 3, 6, 9 and 12 months
  Adherence to Stroke Prevention Medications (Anti platelets, Anticoagulants, Statins, antihypertensives, antidiabetics) measured by Morisky-Green-Levine Adherence Scale (1-4) where higher scores indicate higher levels of reported adherence.
HbA1c | 1, 3, 6, 9 and 12 months
  HbA1c (glycated hemoglobin) value was collected from medical records and recorded as a percentage.
LDL cholesterol | 1, 3, 6, 9 and 12 months
  Low density lipoprotein-cholesterol level was collected from medical records and recorded as mg/dL
Triglyceride | 1, 3, 6, 9 and 12 months
  Triglyceride level was collected from medical records and recorded as mg/dL.
Body mass index | 1, 3, 6, 9 and 12 months
  Body mass index (BMI) was collected from medical records and recorded as kg/m2

SECONDARY OUTCOMES:
Measuring Quality of Life | 3, 6 and 12 months
  The patients' quality of life was evaluated using the Stroke-Specific Quality of Life Scale (SSQOL), and the total quality of life score was calculated, a higher score indicates that the patient has a better quality of life.
The National Institutes of Health Stroke Scale | 24 hours before discharge, 3, 6, 9 and 12 months
  The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS), is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid in planning post-acute care disposition.
Stroke Recurrence | 1 year
  Stroke recurrence (radiologically and clinically confirmed) within 1 year
Drug Related Problem | 1 year
  Determination of drug-related problems (DRP) using Pharmaceutical Care Network Europe (PCNE) Version 9.1. The basic classification has 3 primary domains for problems, 9 primary domains for causes and 5 primary domains for Planned Interventions, 3 primary domains for level of acceptance (of interventions) and 4 primary domains for the Status of the problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cengiz KN, Midi I, Sancar M. The effect of clinical pharmacist-led pharmaceutical care services on medication adherence, clinical outcomes and quality of life in patients with stroke: a randomised controlled trial. Int J Clin Pharm. 2025 Feb;47(1):99-106. doi: 10.1007/s11096-024-01811-0. Epub 2024 Oct 12. PMID 39395139